CLINICAL TRIAL: NCT02695797
Title: Immunotherapy in Intractable Cryptogenic Epilepsy Patients With Autoimmune Antibody
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sang Kun Lee, Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1504102666
Record Dates: First submitted 2015-06-18; First posted 2016-03-01 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Epilepsy, Unspecified, Intractable
Keywords: Intractable cryptogenic epilepsy with autoimmune antibody; Immunotherapy
MeSH Terms: conditions — Epilepsy | interventions — Immunoglobulins, Intravenous; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immunotherapy (Experimental): Intravenous immunoglobulin (IVIG) and oral prednisolone. IVIG and oral prednisolone are administered simultaneously: IVIG (400mg/kg/day for 5 days) with oral prednisolone (60mg for 5days, than decrease by 10 mg every 2 day).
  Interventions: Other: IVIG; Drug: Prednisolone
- Control (No Intervention): No immunotherapy.

INTERVENTIONS:
Other: IVIG — IVIG (400mg/kg/day for 5 days) with oral prednisolone (60mg for 5days, than decrease by 10 mg every 2 day)
  Arms: Immunotherapy
Drug: Prednisolone — IVIG (400mg/kg/day for 5 days) with oral prednisolone (60mg for 5days, than decrease by 10 mg every 2 day)
  Arms: Immunotherapy

SUMMARY:
The purpose of the study is to investigate effect of immunotherapy in intractable cryptogenic epilepsy patients with autoimmune antibody.

DETAILED DESCRIPTION:
Cryptogenic epilepsy is an epilepsy of presumed symptomatic nature but the cause has not been identified. It account for at least 40% of adult-onset epilepsy. Autoimmune encephalitis including classic paraneoplastic syndrome and autoimmune synaptic encephalitis is a new category of immune-mediated disorders which often has favorable outcome. Recent studies reported that immunotherapy improves seizure outcome in medically intractable epilepsy patients with clinical and serological evidence of an autoimmune basis. Neural autoantibodies were detected in 22% of epilepsy due to unknown cause in a study, mostly from the antiepileptic drug(AED)-resistant epilepsy group. Of the patients who received immunotherapy, 75% archived >50% reduction in seizure frequency.

Many patients with cryptogenic epilepsy are refractory to AED and significant percent of cryptogenic epilepsy harbor neural autoantibody. In those cases, immunotherapy is suggestive based on favorable outcome of immunotherapy in autoimmune encephalitis and autoimmune epilepsy. Investigators aim to investigate the response to immunotherapy in intractable cryptogenic epilepsy patients with neural autoantibodies.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of cryptogenic epilepsy according to the International League Against Epilepsy's Classification of Epilepsy.
* Intractable epilepsy: Complete seizure control is not achieved with trials of two appropriate antiepileptic drugs
* At least 1 seizure within the past 8 weeks
* Presence of autoimmune antibody (NMDAR, LGI1, CASPR2, AMPA1, AMPA2, GABAB-R, anti-Hu, -Yo, -Ri, -Ma2, -CV2/CRMP5, -amphiphysin, GAD) in serum or cerebrospinal fluid
* Written informed consent signed by the subject or legal guardian prior to entering the study

Exclusion Criteria:

* Clinical evidence of autoimmune encephalitis such as autoimmune limbic encephalitis
* History of severe head trauma
* Presence of structural abnormality which is thought to be epileptogenic in brain MRI
* Epilepsy of predominantly genetic or presumed genetic origin
* An active CNS infection, demyelinating disease, degenerative neurologic disease or any CNS disease deemed to be progressive during the course of the study that may confound the interpretation of the study results History of immunotherapy
* A history of nonepileptic or psychogenic seizures within past 1 year
* Any clinically significant laboratory abnormality that in the opinion of the Investigator would exclude the subject from the study
* Any clinically significant psychiatric illness, psychological, or behavioral problems that, in the opinion of the Investigator, would interfere with the subject's ability to participate in the study
* Recent (within 4 weeks) change or dose adjustment of anti-epileptic drug (1 to 2 doses of rescue benzodiazepine is permitted)
* Refuse to participate in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Percent seizure reduction | 3 months

SECONDARY OUTCOMES:
Seizure free rate | 3 months
Responder rate | 3 months
Treatment failure rate | 3 months
Quality of life scores as measured by QOLIE-31 | 3 months
Quality of life scores as measured by BDI-2 | 3 months
Cognition scores as measured by K-MMSE | 3 months
Amount of epileptiform discharge measured by EEG | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Sang Kun Lee, Professor, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shorvon SD. The etiologic classification of epilepsy. Epilepsia. 2011 Jun;52(6):1052-7. doi: 10.1111/j.1528-1167.2011.03041.x. Epub 2011 Mar 30. PMID 21449936
- [Background] Dalmau J, Rosenfeld MR. Paraneoplastic syndromes of the CNS. Lancet Neurol. 2008 Apr;7(4):327-40. doi: 10.1016/S1474-4422(08)70060-7. PMID 18339348
- [Background] Dalmau J, Rosenfeld MR. Autoimmune encephalitis update. Neuro Oncol. 2014 Jun;16(6):771-8. doi: 10.1093/neuonc/nou030. Epub 2014 Mar 16. PMID 24637228
- [Background] Shin YW, Lee ST, Shin JW, Moon J, Lim JA, Byun JI, Kim TJ, Lee KJ, Kim YS, Park KI, Jung KH, Lee SK, Chu K. VGKC-complex/LGI1-antibody encephalitis: clinical manifestations and response to immunotherapy. J Neuroimmunol. 2013 Dec 15;265(1-2):75-81. doi: 10.1016/j.jneuroim.2013.10.005. Epub 2013 Oct 17. PMID 24176648
- [Background] Titulaer MJ, McCracken L, Gabilondo I, Armangue T, Glaser C, Iizuka T, Honig LS, Benseler SM, Kawachi I, Martinez-Hernandez E, Aguilar E, Gresa-Arribas N, Ryan-Florance N, Torrents A, Saiz A, Rosenfeld MR, Balice-Gordon R, Graus F, Dalmau J. Treatment and prognostic factors for long-term outcome in patients with anti-NMDA receptor encephalitis: an observational cohort study. Lancet Neurol. 2013 Feb;12(2):157-65. doi: 10.1016/S1474-4422(12)70310-1. Epub 2013 Jan 3. PMID 23290630
- [Background] Lim JA, Lee ST, Jung KH, Kim S, Shin JW, Moon J, Byun JI, Kim TJ, Shin YW, Lee KJ, Kim YS, Park KI, Lee SK, Chu K. Anti-N-methyl-d-aspartate receptor encephalitis in Korea: clinical features, treatment, and outcome. J Clin Neurol. 2014 Apr;10(2):157-61. doi: 10.3988/jcn.2014.10.2.157. Epub 2014 Apr 23. PMID 24829602
- [Background] Kim TJ, Lee ST, Shin JW, Moon J, Lim JA, Byun JI, Shin YW, Lee KJ, Jung KH, Kim YS, Park KI, Chu K, Lee SK. Clinical manifestations and outcomes of the treatment of patients with GABAB encephalitis. J Neuroimmunol. 2014 May 15;270(1-2):45-50. doi: 10.1016/j.jneuroim.2014.02.011. Epub 2014 Feb 28. PMID 24662003
- [Background] Barajas RF, Collins DE, Cha S, Geschwind MD. Adult-onset drug-refractory seizure disorder associated with anti-voltage-gated potassium-channel antibody. Epilepsia. 2010 Mar;51(3):473-7. doi: 10.1111/j.1528-1167.2009.02287.x. Epub 2009 Sep 22. PMID 19780798
- [Background] Majoie HJ, de Baets M, Renier W, Lang B, Vincent A. Antibodies to voltage-gated potassium and calcium channels in epilepsy. Epilepsy Res. 2006 Oct;71(2-3):135-41. doi: 10.1016/j.eplepsyres.2006.06.003. Epub 2006 Jul 25. PMID 16870397
- [Background] Liimatainen S, Peltola M, Sabater L, Fallah M, Kharazmi E, Haapala AM, Dastidar P, Knip M, Saiz A, Peltola J. Clinical significance of glutamic acid decarboxylase antibodies in patients with epilepsy. Epilepsia. 2010 May;51(5):760-7. doi: 10.1111/j.1528-1167.2009.02325.x. Epub 2009 Oct 8. PMID 19817821
- [Background] Peltola J, Kulmala P, Isojarvi J, Saiz A, Latvala K, Palmio J, Savola K, Knip M, Keranen T, Graus F. Autoantibodies to glutamic acid decarboxylase in patients with therapy-resistant epilepsy. Neurology. 2000 Jul 12;55(1):46-50. doi: 10.1212/wnl.55.1.46. PMID 10891904
- [Background] Bien CG. Value of autoantibodies for prediction of treatment response in patients with autoimmune epilepsy: review of the literature and suggestions for clinical management. Epilepsia. 2013 May;54 Suppl 2:48-55. doi: 10.1111/epi.12184. PMID 23646971
- [Background] Toledano M, Britton JW, McKeon A, Shin C, Lennon VA, Quek AM, So E, Worrell GA, Cascino GD, Klein CJ, Lagerlund TD, Wirrell EC, Nickels KC, Pittock SJ. Utility of an immunotherapy trial in evaluating patients with presumed autoimmune epilepsy. Neurology. 2014 May 6;82(18):1578-86. doi: 10.1212/WNL.0000000000000383. Epub 2014 Apr 4. PMID 24706013
- [Background] Brenner T, Sills GJ, Hart Y, Howell S, Waters P, Brodie MJ, Vincent A, Lang B. Prevalence of neurologic autoantibodies in cohorts of patients with new and established epilepsy. Epilepsia. 2013 Jun;54(6):1028-35. doi: 10.1111/epi.12127. Epub 2013 Mar 6. PMID 23464826
- [Background] Iorio R, Assenza G, Tombini M, Colicchio G, Della Marca G, Benvenga A, Damato V, Rossini PM, Vollono C, Plantone D, Marti A, Batocchi AP, Evoli A. The detection of neural autoantibodies in patients with antiepileptic-drug-resistant epilepsy predicts response to immunotherapy. Eur J Neurol. 2015 Jan;22(1):70-8. doi: 10.1111/ene.12529. Epub 2014 Aug 12. PMID 25112548